CLINICAL TRIAL: NCT00206908
Title: BRAIN (Biomarker Rapid Assessment of Ischemic iNjury)
Status: Completed | Type: Observational
Sponsor: Abbott RDx Cardiometabolic (Other)
Other Study IDs: 003
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Stroke; Stroke Mimic(Conditions Presenting With Stroke-like Conditions)
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
This project is designed to evaluate the clinical utility of a novel blood test, the Triage Stroke Panel, as an aid in the diagnosis and assessment of stroke. The Triage Stroke Panel test device, used with the Triage MeterPlus, is a rapid, point-of-care immunoassay. The test measures the concentration of various analytes present in EDTA-anticoagulated whole blood or plasma, specifically B-type natriuretic peptide (BNP), fibrin degradation products containing D-Dimer, matrix metalloproteiase-9 (MMP-9), and S-100B. The test utilizes a proprietary algorithm for the automatic calculation of a single Multimarker Index (MMX) result from the individual biomarker values. The MMX result is being evaluated for use as an aid in the assessment and diagnosis of stroke.

DETAILED DESCRIPTION:
To date, there is no commercially available blood test approved in the United States for use as an aid in the assessment and diagnosis of stroke. There have been various reports in the scientific literature describing the ability of various biomarkers to predict or identify stroke, with varied success. A biomarker panel approach, similar to that used for the evaluation of chest pain patients (troponin I, CK-MB, and myoglobin) enhances diagnostic accuracy, particularly when the panel includes protein markers associated with various components of the disease pathophysiology. This study involves a retrospective analysis of data collected from patients that present with an acute focal neurological deficit, suspected cerebral ischemia, or suspected intracranial hemorrhage within 24 hours of symptom onset or last known well time will be enrolled into the study. Blood samples will be collected at enrollment and serially up to 72 hrs. from the time of onset or last known well time. The study population will also include a subset of patients with subarachnoid hemorrhage, who will have additional samples collected daily from day 3 through day 14 (at clinical sites participating in the vasospasm substudy) for the evaluation of cerebral vasospasm. The patient's participation in the study is complete when all samples have been collected or when they are discharged from the hospital, whichever occurs first. All blood sample will be analyzed using the Triage Stroke Panel test. Measurements will be performed at each clinical site and at Biosite (subject to test device availability). In order to minimize bias and eliminate significant risk to the patient, physicians will be blinded to all Triage Stroke Panel results during the course of the study. Completed case report forms (CRFs) and frozen plasma samples will be transferred to Biosite.

ELIGIBILITY:
Inclusion Criteria:

Age 18 and above Cerebral ischemia or intracranial hemorrhage suspected Enrollment within 24 hrs from symptom onset or last well-known time

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cerebral ischemia or intracranial hemorrhage suspected.
Sampling Method: Probability Sample
Enrollment: 900
Dates: Start 2002-07

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Laskowitz, MD, Principal Investigator — Duke University Hospital
Locations (22):
- United States (18):
  - Alabama Neurological Institute, Birmingham, Alabama
  - University of California, Los Angeles Medical Center, Los Angeles, California
  - Denver Health, Denver, Colorado
  - University of Colorado Health Science Center, Denver, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Kentucky Neuroscience Research, Louisville, Kentucky
  - University of Massachusettes, Worcester Medical Center, Worcester, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Ingham Regional Medical Center, Lansing, Michigan
  - Henepin County Medical Center, Minneapolis, Minnesota
  - St. Luke's Health System, Kansas City, Missouri
  - Duke University Hopsital, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Hospital at the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Sentara Norfolk General Hospital, Norfolk, Virginia
- Toronto Western Hospital, Toronto, Ontario, Canada
- Neurologische Universitatsklinik/Heidelberg, Heidelberg, Germany
- CHUV-Lausanne, Lausanne, Switzerland
- University of Nottingham, Nottingham, United Kingdom